CLINICAL TRIAL: NCT03227120
Title: The Effects of Prehabilitative Exercise on Functional Recovery Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Radford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#2242
Record Dates: First submitted 2017-05-15; First posted 2017-07-24 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Arthroplasty; Osteoarthritis, Knee
Keywords: Exercise Therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial with repeated measures pre and post-surgery. Consecutive patients which meet inclusion and exclusion criteria and consent to participate will be evaluated two months or more pre-operatively. After completion of office testing at the pre-surgery/pre-exercise time point, randomization will be completed using a gender stratified randomized sequence generated prior to subject recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Exercise (Experimental): Receives Prehabilitation exercise program for three times a week for eight weeks of direct outpatient exercise instruction.
  Interventions: Other: Prehabilitation exercise
- Control (No Intervention): Receives the usual standard of care which is a one time Strength and Flexibility written home exercise program provided during total joint education pre-surgery class.

INTERVENTIONS:
Other: Prehabilitation exercise — Three times weekly exercise program of strengthening, balance and functional activities.
  Weekly evaluation and progression with daily use of the Borg Rating of Perceived Exertion (RPE) supplemented with Heart Rate (HR) and Blood Pressure as needed to target the moderate intensity training level (40-60% HR Max) or above as appropriate to each individual.
  Arms: Prehabilitation Exercise

SUMMARY:
The primary aim of this study is to determine the effects of pre-surgery exercise known as Prehabilitation, on functional outcomes for patients following Total Knee Arthroplasty (TKA) surgery. The hypothesis is patients that receive effective pre-surgery prehabilitation will demonstrate improved recovery as measured by the 6-minute walk (6MW) test at one month post surgery.

DETAILED DESCRIPTION:
People with knee arthritis have lower levels of physical activity and are more susceptible to suffer from additional medical conditions of heart disease, respiratory conditions, diabetes and stroke. For patients with end stage knee osteoarthritis, total knee arthroplasty (TKA) has been widely accepted as beneficial for increased patient satisfaction and improved function. To provide high quality of care and optimize TKA outcomes, healthcare providers need to make decisions about resource allocation. The theory of Prehabilitation proposes to increase strength, balance and endurance prior to surgery with the benefit of less decline and improved rate of recovery following surgery. Preoperative quadriceps strength and walking ability have been shown to be predictive of function one year post operation. However, systematic reviews of Prehabilitation have been inconclusive and this warrants additional investigation.

Prior studies of Prehabilitation have been inadequately designed or have low levels of therapeutic validity. A prior study completed in Spain provided pre-surgical exercise three times weekly for eight weeks and provides an example of high therapeutic validity with the corresponding significant results post-operation. The objective of this study is to translate knowledge of the pre-surgical exercise program completed in Spain into the local context of a hospital system in Virginia. Due to local area considerations of equipment and time, modifications of the Spanish pre-surgical exercise program are to be tested. These adaptations will allow for implementation within American College of Sports Medicine strength training guidelines using individualized exercise progressions and completion of three clinic based sessions per week.

Subjects that provide informed consent and complete initial screening will be scheduled for two pre-surgical and two post-surgical assessment sessions. On the first assessment session, subjects will be classified into three levels adapted from prior research and input from clinicians and administration to determine the need for pre-surgical preparation. Those subjects in the two most severe levels will be asked to participate in a Prehabilitation exercise program for three times a week for eight weeks and if consent is provided, will be randomized into the control (Joint Education Home Exercise Class only) or the intervention exercise program using a gender stratified randomized sequence generated prior to subject recruitment. The researcher will notify sequential subjects of their group allocation based on the predetermined randomized sequence at the end of the first testing session.

The goal of the prehabilitative exercise is to provide an individualized exercise program to be completed 3x/week for 8 weeks. The exercise sessions will be completed in the rehabilitation office at the Institute of Orthopedics and Neurology (ION) by physical therapy students with oversight from licensed PT at no cost for each subject. Ongoing evaluation of each exercise session will use the Borg Rating of Perceived Exertion (RPE) supplemented with Heart Rate (HR) and Blood Pressure as needed to target the moderate intensity training level (40-60% HR Max) or above as appropriate to each individual. Weekly evaluation of each individual's exercise program will be completed and progressed as able. Outline of Exercise program includes:

* Warm-up (Low intensity < 40% HR Max) 5 minutes of walking or bike
* Flexibility: knee flexion/ext and hamstring stretching
* Strengthening, Balance and Functional activities (Moderate intensity 40-60% HR Max)

  o Closed kinetic chain exercises for balance and strengthening: 2-3 sets of 8-20 reps
  * Calf raises unilateral/bilateral
  * Quarter squats progressed to full squats as tolerated
  * Resisted Step Progression (goal of isolated quads)
* Lunge with and without upper extremity support
* Step-ups anteriorly
* Step-downs laterally

  ▪ Balance program (goal of Single Leg Stance (SLS) and BOSU wobble board unilateral for 30 seconds)
* Weight shifts L/R and A/P
* Standing marching
* Single leg stance
* BOSU B maintain stability
* BOSU B with R/L rocking, A/P rocking
* BOSU B with quarter squats
* BOSU Unilateral

  o Progressive Resistance exercises with elastic resistance bands 3 sets of 8-12 RM with 2 min rest period between sets:
  * Leg Press bilateral to unilateral (alternate use of total gym or resisted squats)
  * Seated Knee Extensions
  * Standing Knee Curls
  * Elastic band resisted hip ABD L/R (start with side-lying resisted clam shells)
* Manual therapy according to individual patient needs using a pragmatic approach to assist with weight bearing activity (for example squats)
* Cool-down 5 minutes (Low intensity < 40% HR Max) of walking or bike

Statistical comparisons will be conducted using a repeated measures linear mixed model with group, time and group by time as independent variables. Analyses will be adjusted for age, gender, BMI and baseline of the outcome measure. The primary outcome will be the 6MW pre-surgery/pre-exercise compared to one month post-surgery. Secondary outcomes include relevant clinical metrics (e.g. acute length of stay), impairment measures (e.g. strength), physical performance tests (e.g. gait speed and the six-minute walk test), physical activity measured by Actigraph accelerometer, and patient reported outcomes (e.g. PROMIS for global health). All measures will be collected at four time points:

T1) approximately twelve weeks pre-surgery & before starting the exercise program; T2) approximately two weeks pre-surgery & after completion of the exercise program; T3) one month after joint replacement surgery; and T4) three months after joint replacement surgery.

Potential benefits at the individual level include improved recovery of function post TKA, and improved overall physical activity. Potential benefits at the company/societal level are improved surgical rehabilitation outcomes including shorter hospital stay, quicker return to function, and decreased pain. In addition, collaboration between the orthopedists, physical therapists and administration to implement new methods such as Prehabilitation contribute to meeting the triple aim of healthcare of improved customer service, higher quality and cost savings as required by Medicare payment bundling.

ELIGIBILITY:
Inclusion Criteria:

* waiting on primary unilateral Total Knee Arthroplasty for knee osteoarthritis
* agree to participate including completion of a guided exercise program three times per week for eight weeks

Exclusion Criteria:

* current tobacco use,
* body mass index (BMI) greater than 40 kg/m2,
* pain present in the contralateral limb of 5/10 or more during stair climbing,
* knee or hip replacement surgery in the previous year.
* any medical conditions for which moderate or vigorous exercise is contraindicated. For example uncontrolled stage 2 or 3 hypertension risk group B or C (Pescatello 2004)
* any disease that severely effects functional performance. For example Stroke or Parkinson's disease.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change of Six-minute walk test over time | Six months: from baseline through completion of the study at approximately three months after surgery
  Assesses distance walked over six minutes at a preferred walking speed

SECONDARY OUTCOMES:
Change of Manual muscle tests of hip flexion, extension, abduction; knee flexion, extension and ankle dorsiflexion over time | Average of six months: from baseline through completion of the study at approximately three months after surgery
  Standard muscle testing positions quantified using the MicroFET2
Change of Knee Injury and Osteoarthritis Outcome Score (KOOS) over time | Average of six months: from baseline through completion of the study at approximately three months after surgery
  Self-reported outcome questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: William H Kolb, DPT, Principal Investigator — Radford University
Locations (1):
- Institute for Orthopaedics and Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) will be de-identified. All IPD will only be available to members of the research team and stored on a Carilion password protected computer and protected drive. Any data for analysis will be de-identified and only the minimum required for analysis will be provided.
Supporting Information: Study Protocol
Time Frame: December 2019 or 6 months after the final subject data has been recorded
Access Criteria: Data which have been de-identified will be shared only within the research team.

REFERENCES:
- [Background] Artz N, Elvers KT, Lowe CM, Sackley C, Jepson P, Beswick AD. Effectiveness of physiotherapy exercise following total knee replacement: systematic review and meta-analysis. BMC Musculoskelet Disord. 2015 Feb 7;16:15. doi: 10.1186/s12891-015-0469-6. PMID 25886975
- [Background] Bade MJ, Kohrt WM, Stevens-Lapsley JE. Outcomes before and after total knee arthroplasty compared to healthy adults. J Orthop Sports Phys Ther. 2010 Sep;40(9):559-67. doi: 10.2519/jospt.2010.3317. PMID 20710093
- [Background] Bade MJ, Wolfe P, Zeni JA, Stevens-Lapsley JE, Snyder-Mackler L. Predicting poor physical performance after total knee arthroplasty. J Orthop Res. 2012 Nov;30(11):1805-10. doi: 10.1002/jor.22140. Epub 2012 Apr 26. PMID 22539338
- [Background] Bade MJ, Struessel T, Dayton M, Foran J, Kim RH, Miner T, Wolfe P, Kohrt WM, Dennis D, Stevens-Lapsley JE. Early High-Intensity Versus Low-Intensity Rehabilitation After Total Knee Arthroplasty: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Sep;69(9):1360-1368. doi: 10.1002/acr.23139. Epub 2017 Aug 13. PMID 27813347
- [Background] Barbay K. Research evidence for the use of preoperative exercise in patients preparing for total hip or total knee arthroplasty. Orthop Nurs. 2009 May-Jun;28(3):127-33. doi: 10.1097/NOR.0b013e3181a46a09. PMID 19494760
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Calatayud J, Casana J, Ezzatvar Y, Jakobsen MD, Sundstrup E, Andersen LL. High-intensity preoperative training improves physical and functional recovery in the early post-operative periods after total knee arthroplasty: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Sep;25(9):2864-2872. doi: 10.1007/s00167-016-3985-5. Epub 2016 Jan 14. PMID 26768606
- [Background] Cabilan CJ, Hines S, Munday J. The effectiveness of prehabilitation or preoperative exercise for surgical patients: a systematic review. JBI Database System Rev Implement Rep. 2015 Jan;13(1):146-87. doi: 10.11124/jbisrir-2015-1885. PMID 26447015
- [Background] Caracciolo B, Giaquinto S. Determinants of the subjective functional outcome of total joint arthroplasty. Arch Gerontol Geriatr. 2005 Sep-Oct;41(2):169-76. doi: 10.1016/j.archger.2005.01.005. Epub 2005 Mar 21. PMID 16085068
- [Background] Coudeyre E, Jardin C, Givron P, Ribinik P, Revel M, Rannou F. Could preoperative rehabilitation modify postoperative outcomes after total hip and knee arthroplasty? Elaboration of French clinical practice guidelines. Ann Readapt Med Phys. 2007 Apr;50(3):189-97. doi: 10.1016/j.annrmp.2007.02.002. Epub 2007 Feb 15. PMID 17343953
- [Background] Desmeules F, Hall J, Woodhouse LJ. Prehabilitation improves physical function of individuals with severe disability from hip or knee osteoarthritis. Physiother Can. 2013 Spring;65(2):116-24. doi: 10.3138/ptc.2011-60. PMID 24403671
- [Background] Durrand JW, Batterham AM, Danjoux GR. Pre-habilitation. I: aggregation of marginal gains. Anaesthesia. 2014 May;69(5):403-6. doi: 10.1111/anae.12666. No abstract available. PMID 24738795
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Harding P, Holland AE, Delany C, Hinman RS. Do activity levels increase after total hip and knee arthroplasty? Clin Orthop Relat Res. 2014 May;472(5):1502-11. doi: 10.1007/s11999-013-3427-3. Epub 2013 Dec 19. PMID 24353051
- [Background] Hoogeboom TJ, Oosting E, Vriezekolk JE, Veenhof C, Siemonsma PC, de Bie RA, van den Ende CH, van Meeteren NL. Therapeutic validity and effectiveness of preoperative exercise on functional recovery after joint replacement: a systematic review and meta-analysis. PLoS One. 2012;7(5):e38031. doi: 10.1371/journal.pone.0038031. Epub 2012 May 31. PMID 22675429
- [Background] Kennedy DM, Stratford PW, Riddle DL, Hanna SE, Gollish JD. Assessing recovery and establishing prognosis following total knee arthroplasty. Phys Ther. 2008 Jan;88(1):22-32. doi: 10.2522/ptj.20070051. Epub 2007 Nov 6. PMID 17986495
- [Background] McGinn TG, Guyatt GH, Wyer PC, Naylor CD, Stiell IG, Richardson WS. Users' guides to the medical literature: XXII: how to use articles about clinical decision rules. Evidence-Based Medicine Working Group. JAMA. 2000 Jul 5;284(1):79-84. doi: 10.1001/jama.284.1.79. PMID 10872017
- [Background] Mistry JB, Elmallah RD, Bhave A, Chughtai M, Cherian JJ, McGinn T, Harwin SF, Mont MA. Rehabilitative Guidelines after Total Knee Arthroplasty: A Review. J Knee Surg. 2016 Apr;29(3):201-17. doi: 10.1055/s-0036-1579670. Epub 2016 Mar 10. PMID 26963074
- [Background] Mizner RL, Petterson SC, Stevens JE, Axe MJ, Snyder-Mackler L. Preoperative quadriceps strength predicts functional ability one year after total knee arthroplasty. J Rheumatol. 2005 Aug;32(8):1533-9. PMID 16078331
- [Background] Mizner RL, Petterson SC, Clements KE, Zeni JA Jr, Irrgang JJ, Snyder-Mackler L. Measuring functional improvement after total knee arthroplasty requires both performance-based and patient-report assessments: a longitudinal analysis of outcomes. J Arthroplasty. 2011 Aug;26(5):728-37. doi: 10.1016/j.arth.2010.06.004. Epub 2010 Sep 20. PMID 20851566
- [Background] Murphy L, Helmick CG. The impact of osteoarthritis in the United States: a population-health perspective. Am J Nurs. 2012 Mar;112(3 Suppl 1):S13-9. doi: 10.1097/01.NAJ.0000412646.80054.21. PMID 22373741
- [Background] Oatis CA, Li W, DiRusso JM, Hoover MJ, Johnston KK, Butz MK, Phillips AL, Nanovic KM, Cummings EC, Rosal MC, Ayers DC, Franklin PD. Variations in Delivery and Exercise Content of Physical Therapy Rehabilitation Following Total Knee Replacement Surgery: A Cross-Sectional Observation Study. Int J Phys Med Rehabil. 2014;Suppl 5:002. doi: 10.4172/2329-9096.S5-002. Epub 2014 Apr 22. PMID 26594649
- [Background] Paxton RJ, Melanson EL, Stevens-Lapsley JE, Christiansen CL. Physical activity after total knee arthroplasty: A critical review. World J Orthop. 2015 Sep 18;6(8):614-22. doi: 10.5312/wjo.v6.i8.614. eCollection 2015 Sep 18. PMID 26396937
- [Background] Pescatello LS, Franklin BA, Fagard R, Farquhar WB, Kelley GA, Ray CA; American College of Sports Medicine. American College of Sports Medicine position stand. Exercise and hypertension. Med Sci Sports Exerc. 2004 Mar;36(3):533-53. doi: 10.1249/01.mss.0000115224.88514.3a. PMID 15076798
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Rosenberg N, Nierenberg G, Lenger R, Soudry M. Walking ability following knee arthroplasty: a prospective pilot study of factors affecting the maximal walking distance in 18 patients before and 6 months after total knee arthroplasty. Knee. 2007 Dec;14(6):489-92. doi: 10.1016/j.knee.2007.07.010. Epub 2007 Sep 4. PMID 17766122
- [Background] Silva M, Shepherd EF, Jackson WO, Pratt JA, McClung CD, Schmalzried TP. Knee strength after total knee arthroplasty. J Arthroplasty. 2003 Aug;18(5):605-11. doi: 10.1016/s0883-5403(03)00191-8. PMID 12934213
- [Background] Singh JA, Lewallen DG. Patient-level improvements in pain and activities of daily living after total knee arthroplasty. Rheumatology (Oxford). 2014 Feb;53(2):313-20. doi: 10.1093/rheumatology/ket325. Epub 2013 Oct 25. PMID 24162150
- [Background] Snow R, Granata J, Ruhil AV, Vogel K, McShane M, Wasielewski R. Associations between preoperative physical therapy and post-acute care utilization patterns and cost in total joint replacement. J Bone Joint Surg Am. 2014 Oct 1;96(19):e165. doi: 10.2106/JBJS.M.01285. PMID 25274793
- [Background] Stevens JE, Mizner RL, Snyder-Mackler L. Quadriceps strength and volitional activation before and after total knee arthroplasty for osteoarthritis. J Orthop Res. 2003 Sep;21(5):775-9. doi: 10.1016/S0736-0266(03)00052-4. PMID 12919862
- [Background] Swank AM, Kachelman JB, Bibeau W, Quesada PM, Nyland J, Malkani A, Topp RV. Prehabilitation before total knee arthroplasty increases strength and function in older adults with severe osteoarthritis. J Strength Cond Res. 2011 Feb;25(2):318-25. doi: 10.1519/JSC.0b013e318202e431. PMID 21217530
- [Background] Valkenet K, van de Port IG, Dronkers JJ, de Vries WR, Lindeman E, Backx FJ. The effects of preoperative exercise therapy on postoperative outcome: a systematic review. Clin Rehabil. 2011 Feb;25(2):99-111. doi: 10.1177/0269215510380830. Epub 2010 Nov 8. PMID 21059667
- [Background] Wang L, Lee M, Zhang Z, Moodie J, Cheng D, Martin J. Does preoperative rehabilitation for patients planning to undergo joint replacement surgery improve outcomes? A systematic review and meta-analysis of randomised controlled trials. BMJ Open. 2016 Feb 2;6(2):e009857. doi: 10.1136/bmjopen-2015-009857. PMID 26839013
- [Background] Walsh M, Woodhouse LJ, Thomas SG, Finch E. Physical impairments and functional limitations: a comparison of individuals 1 year after total knee arthroplasty with control subjects. Phys Ther. 1998 Mar;78(3):248-58. doi: 10.1093/ptj/78.3.248. PMID 9520970
- [Background] Waugh EJ, Badley EM, Borkhoff CM, Croxford R, Davis AM, Dunn S, Gignac MA, Jaglal SB, Sale J, Hawker GA. Primary care physicians' perceptions about and confidence in deciding which patients to refer for total joint arthroplasty of the hip and knee. Osteoarthritis Cartilage. 2016 Mar;24(3):451-7. doi: 10.1016/j.joca.2015.09.017. Epub 2015 Oct 23. PMID 26432986
- See also: Center for Disease Control numbers of joint replacements per year — http://www.cdc.gov/nchs/data/databriefs/db210.htm.